CLINICAL TRIAL: NCT04629495
Title: Rapamycin - Effects on Alzheimer's and Cognitive Health (REACH)
Brief Title: Rapamycin - Effects on Alzheimer's and Cognitive Health
Acronym: REACH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC20200763H
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
Keywords: Cognition; Alzheimer's disease biomarkers; Neuroimaging
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: placebo controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RAPA (rapamycin) treatment group (Active Comparator): Subjects will receive active drug
  Interventions: Drug: Rapamycin
- Placebo group (Placebo Comparator): Subjects will receive placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rapamycin — RAPA will be administered orally 1mg daily
  Other Names: Sirolimus, RAPA
  Arms: RAPA (rapamycin) treatment group
Other: Placebo — Placebo will be administered orally once daily
  Other Names: Placebo capsule
  Arms: Placebo group

SUMMARY:
This study will evaluate the safety, tolerability, and feasibility of 12 month oral rapamycin treatment in older adults with amnestic mild cognitive impairment (aMCI) and early stage Alzheimer's disease (AD).

DETAILED DESCRIPTION:
The study will consist of a screening/baseline period of up to 90 days pre-study drug, with a 12-month (+3 day) treatment period with rapamycin, followed by a post-treatment assessment completed within 14 days of the final study drug dose, and a final assessment conducted 6-months (+14 days) after the final study drug dose. The study duration is not expected to exceed 90 weeks for participants.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders and all ethnic groups
2. Ages 55 to 89 years
3. Diagnosis of MCI or AD (Mini Mental Status Examination (MMSE): 18-30; Clinical Dementia Rating Scale (CDR) = 0.5 - 1; California Verbal Learning Test III (CVLT-III) Delayed Recall ≤16% based on age-adjusted norms, clinician approval)
4. Amyloid positivity based on Amyloid PET Imaging
5. Labs: Normal blood cell counts without clinically significant excursions; normal liver and renal function; and glucose control (HbA1c < 6.5%). Fasting lipid panel and prothrombin time/prothrombin time test/international normalized ration (PT/PTT/INR) within normal limits
6. A legally authorized representative (LAR) designated to sign informed consent (if necessary) must attend the Screening visit and accompany the participant to all remaining visits to provide reported outcomes
7. Stable dose of AD medications (Donepezil, rivastigmine, Memantine, galantamine) for at least three months is allowed

Exclusion Criteria:

1. Diabetes (HBA1c≥6.5% or antidiabetic medications)
2. History of skin ulcers or poor wound healing
3. Current tobacco or illicit drug use or alcohol abuse
4. Use of anti-platelet or anti-coagulant medications other than aspirin
5. Current medications that affect cytochrome 450 3A4 (CYP3A4)
6. Immunosuppressant therapy within the last year
7. Chemotherapy or radiation treatment within the last year
8. Current or chronic history of liver or kidney disease or known hepatic or biliary abnormalities
9. Untreated hypertriglyceridemia (fasting triglycerides < 250 mg/dl)
10. Current or chronic history of pulmonary disease or abnormal pulse oximetry (<90%)
11. Chronic heart failure
12. Pregnancy or lactation
13. Recent history (past six months) of myocardial infarction, active coronary artery disease, intestinal disorders, stroke, or transient ischemic attack
14. Significant neurological conditions other than AD or MCI
15. Poorly controlled blood pressure (systolic BP>160, diastolic BP>90 mmHg - based on two readings)
16. Active inflammatory, COVID-19, autoimmune, infectious, hepatic, gastrointestinal, malignant, and/or severe mental illness
17. History of, or MRI, or CT positive for, any space occupying lesion, including mass effect or abnormal intracranial pressure, which would indicate contraindications to lumbar puncture
18. Organ transplant recipients

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events | Baseline to 12 months
  Development or worsening of medical symptoms or problems
Change in glucose level | Baseline to 12 months
  A comprehensive metabolic panel is used to measure change in glucose level
Change in albumin | Baseline to 12 months
  A comprehensive metabolic panel is used to measure change in albumin level
Change in carbon dioxide or bicarbonate (CO2) | Baseline to 12 months
  A comprehensive metabolic panel is used to measure change in CO2
Change in calcium | Baseline to 12 months
  A comprehensive metabolic panel is used to measure change in calcium levels

SECONDARY OUTCOMES:
Central nervous system penetration of rapamycin | Baseline and 12 months
  A lumbar puncture and blood draw will be used to evaluate levels of study drug
Change in Cognition using preclinical Alzheimer's Cognitive Composite 5 (PACC5) | Baseline to 12 months
  Cognition will be measured using the PACC5 scale. The PACC5 is a composite score comprised of measures of global cognition, memory, and executive function. The score reflects an averaged z-score. Scores range from -3 to +3 with higher scores indicating better cognitive performance.
Change in Cognition using Clinical Dementia Rating Scale sum of Boxes (CDR-SOB) | Baseline to 12 months
  CDR is obtained through semistructured interviews of patients and informants, and cognitive functioning is rated in 6 domains of functioning: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Each domain is rated on a 5-point scale of functioning as follows: 0, no impairment; 0.5, questionable impairment; 1, mild impairment; 2, moderate impairment; and 3, severe impairment. Domain scores are entered into an online algorithm and CDR-SOB score obtained by summing each of the domain box scores, ranging from 0 to 18. A lower score indicates better cognition.
Change in Functional status | Baseline to 12 months
  Functional status will be measured using the functional assessment scale (FAS). The FAS is completed by a collateral source and assesses ability to complete instrumental activities of daily living. The scale has 10-items and responses range from 0-3. The total score is a sum of the individual items. The total score ranges from 0 to 30 with higher scores indicating more assistance needed.
Change in Neuropsychiatric symptoms | Baseline to 12 months
  Symptoms will be evaluated using the Geriatric Depression Scale 15 Item (GDS-15). The GDS-15 is a self-report questionnaire with 15 items that have response options of 0 or 1. The total score is the sum of the individual items. The total score on the measure ranges between 0 to 15 with higher scores indicating more depressive symptoms.
Change in Gait Speed | Baseline to 12 months
  Gait speed will be evaluated with an electronic gait mat
Change in Grip Strength | Baseline to 12 months
  Grip strength will be evaluated with a hand dynamometer
Change in CSF amyloid beta | Baseline to 12 months
  Cerebrospinal fluid (CSF) levels of amyloid beta
Change in cerebral glucose metabolism | Baseline to 12 months
  Cerebral glucose metabolism is measured using fluorodeoxyglucose-Positron emission tomography (FDG-PET)
Change in Brain Volumetry | Baseline to 12 months
  Measure of brain volumetry using MRI

CONTACTS AND LOCATIONS:
Overall Officials: Sudha J Seshadri, MD, Principal Investigator — UT Health San Antonio
Locations (1):
- Glenn Biggs Institute for Alzheimer's & Neurodegenerative Diseases, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: At study completion
Access Criteria: Through journal publication